CLINICAL TRIAL: NCT05866029
Title: Efficacy of Sequential Denosumab After Teriparatide for 6 Months Compared With Denosumab Monotherapy in Reducing Risk of Osteoporotic Fractures in Patients With New Fractures: a Multicenter Randomized Controlled Trial (STAND Study)
Brief Title: Study of the Key Techniques of Prevention and Treatment of Osteoporotic Refracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-PUMCH-D-006
Record Dates: First submitted 2023-04-28; First posted 2023-05-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Osteoporotic Fractures
Keywords: osteoporosis; osteoporotic fractures; bone turnover markers; imaging biomarkers
MeSH Terms: conditions — Osteoporotic Fractures; Osteoporosis | interventions — Denosumab; Teriparatide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60mg of Denosumab treatment (Active Comparator): Monotherapy with denosumab injection ( 60mg, subcutaneous injection, semi-annually) for 24 months.
  Interventions: Drug: Denosumab
- Teriparatide was sequentially treated with Denosumab (Experimental): 1. Treatment with teriparatide injection ( 20ug, subcutaneous injection, once daily) for 6 months, followed by discontinuation of teriparatide and change to denosumab injection ( 60mg, subcutaneous injection, once every six months) and continued until the 24th month.
  2. Treatment with teriparatide injection ( 20ug, subcutaneous injection, once daily) for 12 months, followed by discontinuation of teriparatide and change to denosumab injection ( 60mg, subcutaneous injection, semi-annually) treatment continued until the 24th month.
  Interventions: Drug: Denosumab; Drug: Teriparatide

INTERVENTIONS:
Drug: Denosumab — Active Comparator: 60mg of Denosumab treatment by subcutaneous injection
Drug: Teriparatide — Teriparatide was sequentially treated with Denosumab
  Arms: Teriparatide was sequentially treated with Denosumab

SUMMARY:
This project anchors osteoporotic fractures, conduct registration and follow-up studies, and conduct prospective treatment studies. By registering for follow-up studies on osteoporotic fractures, it is planned to obtain epidemiological data through registration and follow-up studies; A prospective treatment study for patients with osteoporotic fractures is planned to explore effective treatment strategies through randomized controlled trials; To study biomarkers for osteoporotic refractures, we plan to establish a biomarker warning model through multi omics research; To study imaging biomarkers for osteoporotic refractures, a new imaging technology is proposed to establish an imaging omics warning model.

ELIGIBILITY:
Inclusion Criteria:

1. New brittle hip fractures;
2. New brittle vertebral fractures;
3. New other site fractures and/or total hip or neck of femur or L1-L4 T-value < -1.0;
4. Men or postmenopausal women;
5. Age 45-90 years old;
6. Ability to move autonomously

Exclusion Criteria:

1. bone metabolic diseases except for osteoporosis eg. a. (Osteogenesis Imperfecta, Paget's disease, Osteomalacia), b. Cushing's syndrome, c.hyperprolactinemia;
2. Having primary hyperparathyroidism or hypothyroidism;
3. Had or have osteomyelitis of the jaw or necrosis of the jaw;
4. GFR<30ml/min/1.73m2;
5. Active infection that requires systematic treatment;
6. Used intravenous bisphosphonate, fluoride, or strontium for osteoporosis within 2 years;
7. Used teriparatide and denosumab for osteoporosis within 6 months;
8. Used glucocorticoids (equivalent to >5 mg/day prednisone) for more than 10 days within 6 weeks;
9. The time gap between the first time and the last time oral bisphosphonate for osteoporosis less than 1 year( if used within one year, but the cumulative use is ≤ 1 month, the subject can be enrolled) ;
10. Patients with malignant tumors or bone metastases within 5 years, except tumors that are expected to be cured after treatment;
11. Have hypocalcemia and hypercalcemia;
12. Unexplained elevation of alkaline phosphatase;
13. A serious deficiency of vitamin D (25OHD <10ng/mL);
14. Patients who have previously received external radiation or radiation therapy with bone implants;
15. Uncontrolled comorbidities included heart failure above the New York cardiac Function Scale, glycosylated hemoglobin > 8.5%, and severe arrhythmias;
16. Planned pregnancy and lactation at present or during the study period;
17. Allergic to teriparatide and denosumab;
18. Participating in clinical trials of other drugs at present;
19. subjects do not suitable for this study

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2478 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The main study：The incidence of new vertebral fractures | Within 24 months of treatment
  The main study：the incidence of new vertebral fractures (clinical and imaging) within 24 months of treatment
The sub study：The rate of change in BMD from baseline at lumbar spine in 24 months | Within 24 months of treatment

SECONDARY OUTCOMES:
The main study：New vertebral fractures in 12 months | Within 12 months of treatment
The main study：New hip fractures, new fractures at other sites, and all new fractures at 12 and 24 months | Within 12 months and 24 months of treatment
The main study：The rate of BMD change from the baseline at the lumbar spine, total hip, and femoral neck in 12 and 24 months; | Within 12 months and 24 months of treatment
The main study：The rate of changes from baseline in serum type 1 collagen cross-linked C-terminal peptide (β-CTX) and type 1 procollagen N-terminal propeptide (P1NP) at 6, 12, and 24 months | 6, 12, and 24 months
The main study：The patients' adherence to treatment | 24 months
  Non-adherence rate=Number of patients non-adherencet with teriparatide or denosumab / Total number of patients.
  1. Denosumab Adherence Adherence to denosumab treatment was assessed based on protocol compliance during the study period. Non-adherence was defined as one or more instances in which the scheduled denosumab injection was not administered according to the study protocol, including doses received outside the permissible treatment window (±4 weeks).
  2. Teriparatide Adherence Adherence to teriparatide was evaluated only in the two sequential treatment groups assigned to receive teriparatide. Using patient diary records, non-adherence was defined as an actual-to-expected injection day ratio of less than 80% or greater than 120% over the course of the study period.
The main study：Cost-effectiveness | 24 months
  The incremental cost-effectiveness ratio is defined as the average additional drug cost required per additional fracture event avoided in the intervention group compared to the control group.
The sub study：BMD change at lumbar spine in 12 months | Within 12 months of treatment
The sub study：BMD changes at total hip and femoral neck in 12 and 24 months | Within 12 months and 24 months of treatment
The sub study：Serum β-CTX and P1NP levels at 12 and 24 months | 12 months and 24 months
The sub study：The incidence of new vertebral fractures, hip fractures, new fractures at other sites, and all new fractures in 12 and 24 months | Within 12 months and 24 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Weibo Xia, MD., Study Chair — Peking Union Medical College Hospital
Locations (58):
- China (58):
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Beijing Pinggu Hospital, Beijing
  - Beijing Shijingshan Hospital, Beijing
  - Beijing Yanhua Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Jilin Province FAW General Hospital, Changchun
  - The Second XIANGYA Hospital of Central South University, Changsha
  - Changzhou NO.2 People's Hospital, Changzhou
  - The First People's Hospital of Changzhou, Changzhou
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Fourth Hospital of Sichuan University, Chengdu
  - The Second People's Hospital of Dalian, Dalian
  - Shengli Oilfield Central Hospital, Dongying
  - Affiliated Hospital of Guizhou Medical University, Guiyang
  - Zhejiang Provincial People's Hospital Bijie Hospital, Guizhou
  - The Fourth Hospital of Harbin Medical University, Haerbin
  - The Second Hospital of Jilin University, Haerbin
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital of USTC (Anhui Provincial Hospital), Hefei
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Shandong Provincial Hospital, Jinan
  - The Second Hospital of Shandong University, Jinan
  - Affiliated Hospital of Jining Medical University, Jining
  - Gansu Provincial Hospital, Lanzhou
  - Liaocheng People's Hospital, Liaocheng
  - Jiangxi Provincial People's Hospital, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - Ningbo NO.2 Hospital, Ningbo
  - Qingdao Municipal Hospital, Qingdao
  - Changhai Hospital, Shanghai
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai Sixth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Tongji Hospital of Tongji University, Shanghai
  - Huazhong University of Science and Technology Union Shenzhen Hospital, Shenzhen
  - Shenzhen Shiyan People's Hospital, Shenzhen
  - The Seventh Affiliated Hospital of Sun Yat-sen University, Shenzhen
  - Hebei Medical University Third Hospital, Shijiazhuang
  - Kunshan Hospital of Traditional Chinese Medicine, Suzhou
  - The First People's Hospital of Kunshan, Suzhou
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - First Hospital of Shanxi Medical University, Taiyuan
  - Second Hospital of Shanxi Medical University, Taiyuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Weifang People's Hospital, Weifang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Qinghai University Affiliated Hospital, Xining
  - General Hospital of Ningxia Medical University, Yinchuan
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan
  - Henan Provincial General Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - The Fifth Affiliated Hospital Sun Yat-sen University, Zhuhai
  - PKUCare Luzhong Hospital, Zibo
  - Zibo Central Hospital, Zibo

IPD SHARING:
Plan to Share IPD: Yes
Data related to this study will be made available upon reasonable request.
Supporting Information: Study Protocol